CLINICAL TRIAL: NCT02186782
Title: Concomitant Clomiphene Citrate and Estradiol Versus Clomiphene Citrate Alone in Ovulation Induction: a Randomized Controlled Trial
Brief Title: Concomitant CC and E2 Versus CC Alone in Ovulation Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maher elesawi kamel elesawi (Other)
Responsible Party: Sponsor-Investigator, Maher elesawi kamel elesawi, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ME1
Record Dates: First submitted 2014-06-28; First posted 2014-07-10 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Infertility; Anovulation
Keywords: Clomiphene citrate; Estradiol; Endometrial thickness
MeSH Terms: conditions — Infertility; Anovulation | interventions — Clomiphene; Estradiol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene citrate-Estradiol group (Active Comparator): Women will receive clomiphene citrate and estradiol
  Interventions: Drug: Clomiphene citrate and Estradiol
- Clomiphene citrate group (Active Comparator): Women will receive clomiphene citrate and placebo
  Interventions: Drug: Clomiphene citrate and Placebo

INTERVENTIONS:
Drug: Clomiphene citrate and Estradiol — Women will receive clomiphene citrate (100 mg/day for 5 consecutive days from day 2 of cycle) and estradiol (2 mg/day for 5 consecutive days from day 2 of cycle)
  Other Names: Clomid and Estradiol valerate
  Arms: Clomiphene citrate-Estradiol group
Drug: Clomiphene citrate and Placebo — Women will receive clomiphene citrate (100 mg/day for 5 consecutive days from day 2 of cycle) and placebo (for 5 consecutive days from day 2 of cycle)
  Other Names: Clomid and Placebo
  Arms: Clomiphene citrate group

SUMMARY:
The purpose of this study is to evaluate the effect of concomitant administration of estradiol during use of clomiphene citrate (CC) for induction of ovulation in infertile women.

DETAILED DESCRIPTION:
Women will be randomly divided into two groups; CC-E2 group and CC group. Women in the CC-E2 group will receive CC (100 mg/day for 5 consecutive days from day 2 of cycle) and estradiol (2 mg/day for 5 consecutive days from day 2 of cycle). Women in the CC group will receive CC (100 mg/day for 5 consecutive days from day 2 of cycle) and placebo mimic estradiol (for 5 consecutive days from day 2 of cycle). Transvaginal sonography (TVS) scan will be performed regularly for monitoring of follicular growth (folliculometry); starting from day 10 of the stimulation cycle and repeated every 2-3 days. When there will be at least one follicle ≥ 18 mm in diameter, final oocyte maturation will be induced by intramuscular administration of 10000 IU of human chorionic gonadotropin (HCG) and timed intercourse will be advised. If there will be no follicle ≥ 12 mm by day 16 of the cycle, monitoring of follicular growth will be discontinued and the cycle will be presumed to be anovulatory. Ovulation will be documented by TVS scan one week after triggering of oocyte maturation and will be confirmed by assessing the midluteal serum progesterone level. Each woman will be subjected to ovarian stimulation for a maximum of 3 consecutive cycles except if she gets pregnant in the first or second cycle.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with eugonadotrophic anovulation/oligoovulation.
* Unexplained infertility.

Exclusion Criteria:

* Age < 20 or > 35 years.
* Body mass index (BMI) < 18.5 kg/m2 or > 25 kg/m2.
* Presence of any infertility factor other than anovulation/oligoovulation.
* Previous history of ovarian surgery or surgical removal of one ovary.
* Previous exposure to cytotoxic drugs or pelvic irradiation.
* Metabolic or hormonal abnormalities.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6-8 weeks gestational age
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 6-8 weeks gestational age) divided by the number of women

SECONDARY OUTCOMES:
Endometrial thickness on day of HCG administration | 3 months
  Endometrial thickness by TVS on day of HCG administration

OTHER OUTCOMES:
Ovulation rate | 3 months
  Number of ovulatory cycles divided by the number of stimulation cycles
Number of ovarian follicles ≥ 18 mm on day of HCG administration | 3 months
  Number of ovarian follicles ≥ 18 mm by TVS on day of HCG administration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Badawy, Prof, Principal Investigator — Mansoura University; Maher E Kamel Elesawi, Dr, Study Director — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University
Locations (3):
- Egypt (3):
  - Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private practice settings, Al Mansurah, Dakahlia Governorate
  - Private practice settings, Mīt Ghamr, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: Undecided